CLINICAL TRIAL: NCT04073732
Title: Family Physician Contract Services and Impacts in China Based on Physician Agency Theory
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Hai Fang, Principal Investigator,Professor, Peking University
Other Study IDs: 71774006
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Physician Behavior; Hypertension
Keywords: family physician contract services; physician agency theory; physician Behavior; family physician; health service supply
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- family physician team: Family physician team in four regions (Beijing, Shanghai, Hangzhou and Xia'men), including general practitioners, nurses and public health personnel.

SUMMARY:
In June 2016, the Health Reform Office in the State Council released "the Announcement about Guiding Opinions of Promoting Family Physician Contract Services". Family Physician Contract Service is an important tool to change the health service models in primary care organizations in China. The relationship between patients and physicians can be regarded as principles and agents.

Physician agency theory has been used to study physician behaviors in economics and management. Family physician contract services regulate the principle-agent relationship between patients and physicians using a formal contract, and there are lots of potentials to employ the physician agency theory to study family physician contract services in China. In theoretical aspects, the present project will study the analysis frameworks and methods of family physician contract services in China under the capitation and global budget payment mechanisms after systematically reviewing Chinese and English literatures about the physician agency theory. In empirical aspects, the present project will collect data from family physician contract services and examine the effects of specific contract forms, incentives, and fees on family physician behaviors and their impacts on health status and medical expenditures of hypertensive and diabetic patients.

DETAILED DESCRIPTION:
1. From a theoretical point of view, using the physician agency theory to construct a family physician contract services and a family physician (team) behavior theory analysis framework and research method system suitable for China's national conditions.
2. From the empirical point of view, from the demand side, analyze the needs of the family physician contract service, the status quo, and the behavior of the visit; from the supplier, understand the behavior changes and satisfaction of the family physician (team) after the implementation of the family physician contract service Degree situation
3. From an empirical perspective, from the level of primary medical institutions, use the sample area data to analyze the impact of family physicians' signing services on the number of visits and medical expenses;
4. From an empirical perspective, using the constructed theoretical analysis framework to analyze the implementation of the Chinese family physician contract service, including incentive mechanism (income, incentive performance salary and contract service fee), family physician team composition, family bed service, etc. The impact, especially on the quality and quantity of services.
5. From the empirical point of view, taking the key monitoring population (hypertension patients as an example) as a sample, further study the family physicians' contractual services, the changes in the practice behavior of family physicians to the key monitoring population (hypertension, diabetes patients), health outcomes, medical expenses The effect is to propose policy recommendations for family physicians' contracting services and physicians' behavior in the new medical reform in the future.

ELIGIBILITY:
Inclusion Criteria:

* Family physician

  1. a family doctor (general practitioner), has a formal medical license, does not retire;
  2. must be directly facing the patient, participate in the patient's diagnosis, prescription, treatment and return visits, with the outpatient service as the main treatment;
  3. family doctors average weekly Must receive at least 20 patients and receive an average of no less than 2 days per week;
  4. Signing informed consent.
* Residents 1) Can complete the questionnaire independently； 2）Oral participation.

Exclusion Criteria:

* Family physician Not signing informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1）Family physician team participating in family physician contract services, including family doctors, nurses, public security personnel, etc.; 2) Residents, Residents who come to the community health service center
Sampling Method: Non-Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Number of contracted residents | 2018.1-2019.6
  Health-care quantity
Average treatment time | 2018.1-2019.6
  Health-care quality
Absolute value of diastolic blood pressure | 2018.1-2019.6
  Health outcome
Medical expenses for patients with hypertension | 2018.1-2019.6
  Health-care cost
Number of service residents per day | 2018.1-2019.6
  Health-care quantity
Absolute value of systolic blood pressure | 2018.1-2019.6
  Health outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chiangning District health commission, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Contains a large amount of personal information, this research and various agencies signed a data confidentiality agreement

REFERENCES:
- [Background] Frolich A, Talavera JA, Broadhead P, Dudley RA. A behavioral model of clinician responses to incentives to improve quality. Health Policy. 2007 Jan;80(1):179-93. doi: 10.1016/j.healthpol.2006.03.001. Epub 2006 Apr 19. PMID 16624440
- [Result] Arrow KJ. Uncertainty and the welfare economics of medical care. 1963. Bull World Health Organ. 2004 Feb;82(2):141-9. Epub 2004 Mar 16. No abstract available. PMID 15042238
- [Result] Fang H, Liu H, Rizzo JA. Has the use of physician gatekeepers declined among HMOs? Evidence from the United States. Int J Health Care Finance Econ. 2009 Jun;9(2):183-95. doi: 10.1007/s10754-009-9060-8. Epub 2009 Apr 9. PMID 19357948
- [Result] Fang H, Rizzo JA. Managed care and physicians' perceptions of drug formulary use. Am J Manag Care. 2009 Jun;15(6):395-400. PMID 19514805
- [Result] Wilson DM, Taylor DW, Gilbert JR, Best JA, Lindsay EA, Willms DG, Singer J. A randomized trial of a family physician intervention for smoking cessation. JAMA. 1988 Sep 16;260(11):1570-4. PMID 3411737
- [Result] Avery DM Jr, Hooper DE, McDonald JT Jr, Love MW, Tucker MT, Parton JM. The economic impact of rural family physicians practicing obstetrics. J Am Board Fam Med. 2014 Sep-Oct;27(5):602-10. doi: 10.3122/jabfm.2014.05.140052. PMID 25201930
- [Result] Yip WC, Hsiao W, Meng Q, Chen W, Sun X. Realignment of incentives for health-care providers in China. Lancet. 2010 Mar 27;375(9720):1120-30. doi: 10.1016/S0140-6736(10)60063-3. PMID 20346818
- [Result] Conrad DA. The Theory of Value-Based Payment Incentives and Their Application to Health Care. Health Serv Res. 2015 Dec;50 Suppl 2(Suppl 2):2057-89. doi: 10.1111/1475-6773.12408. Epub 2015 Nov 9. PMID 26549041
- See also: Related Info — http://www.nhc.gov.cn/